CLINICAL TRIAL: NCT03646409
Title: Venous Thromboembolism and Bleeding Risk in Patients With Esophageal Cancer
Acronym: VENETIA
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Harry R. Buller, Prof. dr. H.R. Büller, principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: thromboembolism and bleeding
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Venous Thromboembolism; Esophagus Cancer; Bleeding; Chemotherapy Effect
MeSH Terms: conditions — Venous Thromboembolism; Esophageal Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with esophageal cancer receiving chemotherapy: Patients > 18 years with esophageal cancer receiving neoadjuvant chemotherapy
  Interventions: Other: Venous thromboembolic event, arterial thromboembolic event, bleeding events

INTERVENTIONS:
Other: Venous thromboembolic event, arterial thromboembolic event, bleeding events — Whether or not venous or arterial thromboembolic and bleeding events occur in patients with esophageal cancer receiving neoadjuvant chemotherapy

SUMMARY:
This study aims to assess the 6- and 12-month venous thromboembolism (VTE) and bleeding incidence from the start of cancer diagnosis in a retrospective cohort of patients with esophageal cancer. Additionally, the predictive value of the Khorana score and several other VTE and bleeding prediction scores and risk factors will be evaluated.

DETAILED DESCRIPTION:
Patients with cancer are at high risk of venous thromboembolism (VTE), including deep-vein thrombosis and pulmonary embolism. For cancer patients receiving chemotherapy the incidence of VTE is even higher.

Several predictive models were previously developed to identify and justify thromboprophylaxis for cancer patietns who are at highest risk of VTE, like the Khorana and PROTECHT score. The Khorana score is a risk-stratification tool to select patients at high risk of VTE for thromboprophylaxis. The PROTECHT score takes cisplatin-based chemotherapy into account in addition of the Khorana score.

Thereby, the incidence of bleeding and VTE in patients with esophageal cancer is not clear.

This study aims to assess the 6- and 12-month venous thromboembolism (VTE) and bleeding incidence from the start of cancer diagnosis in a retrospective cohort of patients with esophageal cancer. Additionally, the predictive value of the Khorana score and several other VTE and bleeding prediction scores and risk factors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal cancer patients
* Receiving chemotherapy
* Age at least 18 years old

Exclusion Criteria:

- Death <3 months after cancer diagnosis (baseline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer, receiving chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
VTE- and bleeding incidence | from start of cancer diagnosis
  6- and 12-month VTE- and bleeding incidence

SECONDARY OUTCOMES:
Predictive performance of VTE risk factors and known prediction models | from start cancer diagnosis
  To assess the predictive value of Khorana, modified Vienna-, and PROTECHT score in Predictive performance of VTE risk factors and known prediction models
Predictive performance of bleeding risk factors and known prediction models | from start cancer diagnosis
  Predictive performance of bleeding risk factors and known prediction models
Arterial thromboembolism (ATE) incidence | from start of cancer diagnosis
  6- and 12-month ATE incidence

CONTACTS AND LOCATIONS:
Overall Officials: Harry R Büller, Prof. dr., Principal Investigator — Vascular Medicine
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timp JF, Braekkan SK, Versteeg HH, Cannegieter SC. Epidemiology of cancer-associated venous thrombosis. Blood. 2013 Sep 5;122(10):1712-23. doi: 10.1182/blood-2013-04-460121. Epub 2013 Aug 1. PMID 23908465
- [Background] Khorana AA, Francis CW, Culakova E, Kuderer NM, Lyman GH. Frequency, risk factors, and trends for venous thromboembolism among hospitalized cancer patients. Cancer. 2007 Nov 15;110(10):2339-46. doi: 10.1002/cncr.23062. PMID 17918266
- [Background] Starling N, Rao S, Cunningham D, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR. Thromboembolism in patients with advanced gastroesophageal cancer treated with anthracycline, platinum, and fluoropyrimidine combination chemotherapy: a report from the UK National Cancer Research Institute Upper Gastrointestinal Clinical Studies Group. J Clin Oncol. 2009 Aug 10;27(23):3786-93. doi: 10.1200/JCO.2008.19.4274. Epub 2009 Apr 27. PMID 19398575
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292
- [Background] Pabinger I, Thaler J, Ay C. Biomarkers for prediction of venous thromboembolism in cancer. Blood. 2013 Sep 19;122(12):2011-8. doi: 10.1182/blood-2013-04-460147. Epub 2013 Aug 1. PMID 23908470
- [Background] Verso M, Agnelli G, Barni S, Gasparini G, LaBianca R. A modified Khorana risk assessment score for venous thromboembolism in cancer patients receiving chemotherapy: the Protecht score. Intern Emerg Med. 2012 Jun;7(3):291-2. doi: 10.1007/s11739-012-0784-y. Epub 2012 May 1. No abstract available. PMID 22547369